CLINICAL TRIAL: NCT04662385
Title: The Effect of Toothpaste Containing Aloe Vera on Clinical and Microbiological Out Comes With Measuring IL_1 β in Gingival Crevicular Fluid: a Randomized Controlled Crossover Clinical Trial
Brief Title: The Effect of Toothpaste Containing Aloe Vera on Gingivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zainab J Abbas (Other)
Responsible Party: Sponsor-Investigator, Zainab J Abbas, BCs, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: U0005EDO
Record Dates: First submitted 2020-11-28; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Generalized Gingivitis
MeSH Terms: interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Intervention Model Description: twenty-four adult patients with generalized gingivitis participated in the double blinded randomized controlled crossover study divided into two groups, aloe vera and colgate toothpaste used during seven days , one group received aloe vera toothpaste twice times daily and the second group received colgate toothpaste twice dialy .
Who Masked: Participant, Investigator
Masking Description: third professional person give the one of opaque coded toothpaste to the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aloe vera toothpaste group (Experimental): a recently available aloe vera toothpaste for gingival care, offers a completely improved approach for treatment of gingivitis. aloe vera toothpaste was certified as an antibacterial .This innovative toothgel is made using stabilized aloe vera gel from Forever's own plantations and can help you fight plaque as part of a regular brushing routine.
  Interventions: Drug: aloe vera toothpaste; Drug: Colgate Total
- colegate total toothpaste group (Active Comparator): Active Ingredient: Stannous fluoride 0.454% (0.15% w/v fluoride ion) Purposes: Anticavity, Antigingivitis, Antisensitivity. Inactive ingredients: Zinc phosphate, Water, Sorbitol, Hydrated silica, Glycerin, PEG-12, Tetras
  Interventions: Drug: aloe vera toothpaste; Drug: Colgate Total

INTERVENTIONS:
Drug: aloe vera toothpaste — aloe vera toothpaste have antimicrobial and other multipotential effects.
Drug: Colgate Total — Whitening toothpaste that removes and prevents new stains Fights bacteria on teeth, tongue, cheeks and gums for whole mouth healthy Mint toothpaste for long lasting fresh breath Helps prevent plaque, tartar, cavities & gingivitis
  Other Names: colgate SF

SUMMARY:
Twenty-four adult patients (male and female) with generalized gingivitis participated in the double-blinded randomized crossover trial was divided into two groups, (aloe vera and Colgate toothpaste). a week after receiving polishing and scaling,24hours plaque re-growth, one group received Aloe Vera toothpaste twice times daily and the second group received Colgate toothpaste twice daily. The first visit included PLI measurement after that Investigator removed the supra gingival plaque by cotton roll to avoid contamination with the PERIOPAPER strip during GCF collection, then GCF collected from targeted sites(upper incisors, labial side)and Unstimulated saliva collected (for early colonizer bacterial load S. sanguinis and S. mutant) after that the other clinical periodontal parameters ( BOP) were measured and then scaling was done after sample collection because of gingival bleeding which occur during scaling then inform the patient to use the coded toothpaste which gave to the participant by the assistant not involve in the study so the researcher did not know the type of toothpaste that was given to the participant (Colgate or aloe vera twice daily).The toothpastes was given for one week .The codded toothpaste was gave randomly by a decision on that day for example on Sunday Investigator gave all the participants code 1 and on other days Investigator gave to other participants code 2 .In the second visit the PLI was measured first , then the samples were collected from the same teeth after that the other periodontal parameters were collected again ( BOP). After that, participants entered a 6-day wash out period and they were asked to resume oral hygiene measures. After the washout period, the same protocol was repeated for other type of toothpaste.

DETAILED DESCRIPTION:
One of the most predominant periodontal diseases is the plaque induced gingivitis. Certain plants used in folk medicine serve as a source of therapeutic agents that have antimicrobial and other multipotential effects.

Aim: The aim of study is to evaluate the toothpaste containing high concentration of Aloe Vera on reduction of plaque and gingivitis and on clinical periodontal parameter (PI&BOP) salivary primary colonizers boat (S. sanguinis and S. mutant).and determine the effect of aloe vera toothpaste on the pro inflammatory cytokines (IL_1β) in the gingival crevicular fluid.

Objective To evaluate the efficacy of aloe vera toothpaste on IL_1β by using ELISA technique and evaluate the efficacy of aloe vera toothpaste on early colonizer load using (PCR).

Null hypothesis aloe vera has Anti-Inflammatory effect by reducing IL_1β and some clinical periodontal parameters (plaque index& bleeding on probing index) when used by the patients with regular mechanical oral hygiene.

Alternative hypothesis the effect of aloe vera toothpaste is less than Colgate toothpaste on the inflammatory marker IL_1β, early load and some clinical parameters (PI and BOP).

Materials and methods Twenty-four adult patients (male and female) with generalized gingivitis participated in the double-blinded randomized crossover trial was divided into two groups, (aloe vera and Colgate toothpaste). A week after receiving polishing and scaling,24hours plaque re-growth. In zero day, after 24h and 7 days' time points, plaque index and bleeding on probe was recorded, and then the participants entered a 7-day washout period with regular oral hygiene measures. And 7days to used other type of toothpaste (aloe vera or Colgate).in the first visit (zero day) GCF collected from targeted sites (upper incisors, labial side). In the second visit (after 24 hours) saliva collected (for early colonizer load) and the patient brushing teeth and wait 2 hours, after 2hour saliva collected again. the GCF collected in third visit (after7 days), fourth visit (after wash out period) and fifth visit from the same teeth. Saliva collected in third and fifth visit.

ELIGIBILITY:
Inclusion Criteria:

1) 20_30 years old subject. (2) good general health. (3) presence of more than 20 teeth

-

Exclusion Criteria:

1. active cavity caries and/or periodontal disease.
2. ongoing orthodontic treatment.
3. a history of antibiotics within the past 4 months.
4. require prophylactic antibiotic coverage.
5. require systemic and/or topical non-steroidal anti-inflammatory drugs for the past 4 months.
6. pregnant or intended to and lactating mother.
7. have heart valve replacement and\or any systemic disease.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — twenty-four adult male and female patients with generalized gingivitis
Enrollment: 24 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
measuring interleukin -1 beta | one week
  measure interleukin -1 beta in gingival crevicular fluid by using ELISA
early colonizer load of (S. sanguinis and S. mutant) | one week
  early colonizer load of (S. sanguinis and S. mutant) in saliva by using PCR

SECONDARY OUTCOMES:
measuring plaque accumulation | one week
  measure plaque accumulation on the teeth by measuring the plaque index using disclosing agent (erythrosine tablets).
measure the gingival sulcus erosion | one week
  measure the gingival sulcus erosion and destruction by measuring the bleeding on probing index using periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad university college of dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No